CLINICAL TRIAL: NCT04034368
Title: A Perspective Study of the Antiviral Efficacy and Safety of Switching to TAF Treatment in CHB Adults With Suboptimal Response (SOR) or Intolerant to Entecavir
Brief Title: A Perspective Study of the Antiviral Efficacy and Safety of Switching to TAF Treatment in CHB Adults With Suboptimal Response (SOR) and Intolerant to Entecavir
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yanhang Gao, Professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISR-CN-18-10478
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: HBV
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Arm (Experimental): Tenofovir alafenamide (TAF) 25 mg QD, oral administration, 48 weeks；
  Interventions: Drug: Tenofovir Alafenamide (TAF)

INTERVENTIONS:
Drug: Tenofovir Alafenamide (TAF) — Tenofovir alafenamide (TAF) 25 mg QD, oral administration, 48 weeks；

SUMMARY:
This is a multicenter, single arm, open label, historical control pilot Study to the antiviral efficacy and safety of Suboptimal Responders to Entecavir Switching to TAF Treatment at week 48 (investigate the rates of complete virological response on switching to TAF in patients with Suboptimal response or ETV intolerance to standard ETV= 0.5 mg monotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures;
2. Male and female subjects,18 years of age and older, based on the date of the screening visit;
3. Suboptimal Responders to Entecavir (defined as CHB patients treated with at least 12 months of ETV 0.5mg QD with prior suboptimal response viral load still detectable at week 48).
4. ETV intolerance population (defined as unwilling or poor adherence to administer ETV in fasting food, renal impairment with ETV dosage adjustment required, pts with other unidentified reasons willing to switch, etc);
5. Screening serum ALT level ≤ 10 × ULN;
6. Normal ECG (or if abnormal, determined by the Investigator not to be clinically significant);
7. Must be willing and able to comply with all study requirements.

Exclusion Criteria:

1. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study;
2. Co-infection with HCV, HIV, or HDV;
3. Any history of, or current evidence of, clinical hepatic decompensation (i.e., moderate-severe ascites, encephalopathy or variceal hemorrhage);
4. Evidence of hepatocellular carcinoma (e.g. as evidenced by recent imaging);
5. Abnormal hematological and biochemical parameters, including: Hemoglobin < 10 g/dl, Absolute neutrophil count < 0.75×109/L, Platelets ≤ 50×109/L, AST or ALT > 10 × ULN, Total bilirubin > 2.5 × ULN, Albumin < 3.0 g/dl, INR > 1.5 × ULN;
6. Received solid organ or bone marrow transplant;
7. Recent history of pancreatitis (within 24 weeks prior to the first dose of study medication);
8. Evidence of other autoimmune or metabolic liver diseases (except non-alcoholic fatty liver disease);
9. Significant renal, cardiovascular, pulmonary, or neurological disease in the opinion of the investigator;
10. Malignancy within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection(basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible;
11. Known hypersensitivity to study drugs, metabolites, or formulation excipients;
12. Current alcohol or substance abuse judged by the investigator to potentially interfere with subject compliance;
13. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Main efficacy endpoint | Week 48
  The primary efficacy endpoint is the proportion of subjects with plasma HBV DNA levels below 20 IU/ml at Week 48.

SECONDARY OUTCOMES:
Key secondary efficacy endpoint | Week 24
  The proportion of subjects with plasma HBV DNA < 20 IU/mL at Weeks 24
Key secondary efficacy endpoint | Week 48
  The change from baseline in plasma HBV DNA levels at Weeks 48
Key secondary efficacy endpoint | Week 24 and Week 48
  The proportion of subjects with ALT normalization at Weeks 24 and 48
Key secondary efficacy endpoint | Week 48
  The proportion of subjects with HBeAg seroconversion to anti-HBe at Weeks 48
Key secondary efficacy endpoint | Week 48
  The HBV DNA maintenance rate at week 48 in ETV intolerant pts.
Key secondary efficacy endpoint | Week 48
  The proportion of subjects with HBsAg seroconversion to anti-HBs at Weeks 48
Key secondary efficacy endpoint | Week 48
  The incidence of drug resistant mutations at Weeks 48

IPD SHARING:
Plan to Share IPD: No